CLINICAL TRIAL: NCT03308799
Title: A Randomised, Multicentre, Investigator-Blind, Parallel-Group Trial to Evaluate the Efficacy and Safety of MC2-01 Cream Compared to Vehicle and Active Comparator in Subjects With Mild-to-Moderate Psoriasis Vulgaris
Brief Title: A Clinical Trial Evaluating Efficacy and Safety of MC2-01 Cream
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MC2 Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MC2-01-C2
Record Dates: First submitted 2017-10-09; First posted 2017-10-13 (Actual); Results first posted 2019-10-29 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- MC2-01 Cream (Experimental): MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream. One application daily for 8 weeks
  Interventions: Drug: MC2-01 cream
- Cal/BDP combination (Active Comparator): Calcipotriene/betamethasone (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%). One application daily for 8 weeks.
  Interventions: Drug: Cal/BDP combination
- Cream vehicle (Placebo Comparator): One application daily for 8 weeks.
  Interventions: Drug: Cream vehicle

INTERVENTIONS:
Drug: MC2-01 cream — MC2-01 (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%) cream
  Arms: MC2-01 Cream
Drug: Cal/BDP combination — calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%
  Arms: Cal/BDP combination
Drug: Cream vehicle — Vehicle Cream
  Arms: Cream vehicle

SUMMARY:
This trial is a randomized, investigator-blind, multicentre, vehicle- and comparator-controlled, parallel-group trial with the purpose of evaluating efficacy, safety and convenience of the MC2-01 cream.

DETAILED DESCRIPTION:
The MC2-01 Cream is designed for optimal patient satisfaction - it quickly absorbs into the skin leaving it nicely moisturized allowing patients to move on in daily routines. In this trial, the MC2-01 cream will be compared to a marketed product CAL/BDP combination and vehicle. The purpose of the trial is to compare the clinical efficacy, safety, and convenience of this cream to the marketed product. The trial will include a 8-week treatment period.

ELIGIBILITY:
Inclusion Criteria:

* Provided written informed consent
* Generally healthy males or non-pregnant females, of any race or ethnicity, who are at least 18 years of age at the time of screening
* Have a clinical diagnosis of plaque psoriasis (psoriasis vulgaris) of at least 6 months duration that involves the trunk and/or limbs that is amenable to topical treatment with a maximum of 100 g of trial medication per week
* Have a PGA of disease severity of mild or moderate on the body (trunk and/or limbs)
* An mPASI score of at least 2
* Have a treatment area involving 2- 30% of the body surface area (BSA)

Exclusion Criteria:

* Current diagnosis of unstable forms of psoriasis
* Other inflammatory skin disease in the treatment area that may confound the evaluation of the psoriasis vulgaris
* Presence of pigmentation, extensive scarring, pigmented lesions or sunburn in the treatment areas
* Planned exposure to either natural or artificial sunlight
* History of hypersensitivity to any component of the test product or reference product
* Current or past history of hypercalcemia, vitamin D toxicity, severe renal insufficiency, or severe hepatic disorders
* Systemic treatment with biological therapies
* Use of systemic treatments that suppress the immune system and other systemic chemotherapeutic antineoplastic therapy within 4 weeks prior to the baseline visit and during the trial
* Use of phototherapy within 4 weeks prior to Visit 1/Baseline and during the trial;
* Use of topical treatments, except for emollients and non-medicated shampoos, with a possible effect on psoriasis within 2 weeks prior to Visit 1/Baseline
* Clinical signs of skin infection with bacteria, viruses, or fungi
* Known Human Immunodeficiency Virus (HIV) infection
* Any chronic or acute medical condition that may pose a risk to the safety of the subject, or may interfere with the assessment of safety or efficacy in this trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 794 (Actual)
Dates: Start 2017-10-03 (Actual); Primary Completion 2018-06-08 (Actual); Study Completion 2018-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Linda S. Gold, MD, Principal Investigator — Henry Ford Health System
Locations (3):
- United States (3):
  - Henry Ford Hospital, Detroit, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Richard Herdener, MD, Spokane, Washington

REFERENCES:
- [Derived] Pinter A, Galvan J, Freischlager F. Best Responders and Super-Responders to Calcipotriol and Betamethasone Dipropionate PAD-Cream: A Post Hoc Pooled Analysis of Two Phase 3 Trials. Dermatol Ther (Heidelb). 2025 Jun;15(6):1441-1453. doi: 10.1007/s13555-025-01418-x. Epub 2025 Apr 24. PMID 40274711
- [Derived] Stein Gold L, Pinter A, Armstrong A, Augustin M, Arenberger P, Bhatia N, Praestegaard M, Iversen L, Reich A. Calcipotriene and Betamethasone Dipropionate PAD-Cream Demonstrates Greater Treatment Efficacy in Patients with Moderate-to-Severe Psoriasis Compared to Topical Suspension/Gel: A Subgroup Analysis of Two Phase 3 Studies. Dermatol Ther (Heidelb). 2023 Sep;13(9):2031-2044. doi: 10.1007/s13555-023-00979-z. Epub 2023 Jul 25. PMID 37490268
- [Derived] Feldman SR, Praestegaard M, Andreasen AH, Selmer J, Holm-Larsen T. Validation of the Self-Reported Psoriasis Treatment Convenience Scale (PTCS). Dermatol Ther (Heidelb). 2021 Dec;11(6):2077-2088. doi: 10.1007/s13555-021-00626-5. Epub 2021 Oct 14. PMID 34648147
- [Derived] Stein Gold L, Green LJ, Dhawan S, Vestbjerg B, Praestegaard M, Selmer J. A Phase 3, Randomized Trial Demonstrating the Improved Efficacy and Patient Acceptability of Fixed Dose Calcipotriene and Betamethasone Dipropionate Cream. J Drugs Dermatol. 2021 Apr 1;20(4):420-425. doi: 10.36849/JDD.2021.5653. PMID 33852251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject First Visit: 03-Oct-2017. Last Subject Last Visit: 08-Jun-2018.
Pre-assignment Details: Prior to randomization, the subject entered a washout period (if required) where anti-psoriatic treatment and other relevant medication/treatments were discontinued as defined by the exclusion criteria. The washout/screening period could last for up to 30 days, depending on which disallowed treatments the subject received.
Groups:
- CAL/BDP Combination: CAL/BDP (calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%). One application daily for 8 weeks.
  CAL/BDP combination: calcipotriene/betamethasone dipropionate, w/w 0.005%/0.064%
- Vehicle: One application daily for 8 weeks.
  Vehicle
Period: Overall Study
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Vehicle
Started | 342 | 337 | 115
Completed | 320 | 309 | 94
Not Completed | 22 | 28 | 21

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Vehicle | Total
Number analyzed (Participants) | 342 | 337 | 115 | 794
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.0 (14.4) | 52.6 (13.7) | 50.4 (14.3) | 52.0 (14.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 139 | 116 | 44 | 299
  Male | 203 | 221 | 71 | 495
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 290 | 299 | 102 | 691
  Race: Black or African American | 34 | 20 | 11 | 65
  Race: Asian | 10 | 10 | 1 | 21
  Race: American Indian or Alaska Native | 3 | 3 | 1 | 7
  Race: Native Hawaiian or Other Pacific Islander | 2 | 1 | 0 | 3
  Race: Mutiple | 2 | 3 | 0 | 5
  Race: Other | 1 | 1 | 0 | 2
Region of Enrollment [Number; unit: participants]
  United States | 342 | 337 | 115 | 794
Baseline PGA [Count of Participants; unit: Participants] — Severity of psoriasis at Baseline
  Participants
    Mild psoriasis | 68 | 57 | 20 | 145
    Moderate psoriasis | 274 | 280 | 95 | 649
Baseline mPASI [Mean (Standard Deviation); unit: Calculated score] — The extent and severity of the participant's psoriasis are assessed using a modified PASI scoring system at each 3 areas (arms, trunk and legs) using a scale from 0 - 6. 0 = no psoriasis involvement and 6 = 90-100% involvement.The severity is assessed at each for each of the sign redness, thickness and scaliness using a scale from 0 - 4. 0 represents none and 4 represents very severe.
  Calculated score | 7.3 (3.9) | 7.7 (4.1) | 7.1 (4.1) | 7.4 (4.0)
Baseline BSA [Mean (Standard Deviation); unit: Percentage] — Percentage involvement of psoriasis on the Body Surface Area at Baseline
  Percentage | 7.3 (6.0) | 8.4 (7.0) | 7.5 (6.1) | 7.8 (6.5)
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — Fitzpatrick Skin Type was recorded at baseline using the following classification: I = Pale white skin, blue/hazel eyes, blond/red hair; II = Fair skin, blue eyes; III = Darker white skin; IV = Light brown skin; V = Brown skin; VI = Dark brown or black skin
  Participants
    I | 21 | 21 | 9 | 51
    II | 86 | 88 | 30 | 204
    III | 104 | 112 | 37 | 253
    IV | 87 | 73 | 23 | 183
    V | 30 | 28 | 9 | 67
    VI | 14 | 15 | 7 | 36

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Decrease in the Physicians Global Assessment (PGA) Score of Minimum 2 Points on a Scale From 0-4 From Baseline to Week 8
Description: Psoriasis treatment success rate is measured at week 8 by the use of a Physician Global Assessment (PGA) score. Success is defined as a decrease from Baseline of minimum 2 point on a scale from 0 - 4, where: 0 = Clear; 1 = Almost clear; 2 = Mild Plaque thickening; 3 = Moderate Plaque thickening, 4 = Severe Plaque thickening.
  The number of participants referred in the data sets are the number of participants, who achieved a successful treatment success.
Time Frame: Baseline and 8 weeks
Population: The analysis was based on the PP population.
Measure: Number; unit: Count of participants
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Vehicle
Number analyzed (Participants) | 302 | 279 | 88
Count of participants | 121 | 67 | 4

2. Secondary Outcome: Percentage Change in mPASI Score
Description: The extent and severity of the participant's psoriasis is assessed using a modified PASI scoring system (minus scalp, face, and flexures) at each 3 areas (arms, trunk and legs) using a scale from 0 - 6, where 0 = no psoriasis involvement and 6 = 90-100% involvement.
  The severity is assessed at each 3 areas (arms, trunk and legs) for each of the sign redness, thickness and scaliness using a scale from 0 - 4, where 0 represents none and 4 represents very severe.
  The mPASI score is calculated from the individual scores by use of the following equation:
  Arms 0.2 (Redness + Thickness + Scaliness) E = X Trunk 0.3 (Redness + Thickness + Scaliness) E = Y Legs 0.4 (Redness + Thickness + Scaliness) E = Z
  The sum of X + Y + Z = m-PASI score resulting in a minimum score of 0 and a maximum score (worst possible) of 64.8.
  The percent change in mPASI score is defined as the Baseline minus the Week 8 divided by Baseline score multiplied by 100
Time Frame: Baseline and 8 weeks
Population: The analysis was based on the PP population.
Measure: Mean (Standard Deviation); unit: Percentage of change
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Vehicle
Number analyzed (Participants) | 302 | 279 | 88
Percentage of change | 64.8 (28.7) | 52.3 (33.3) | 25.7 (35.3)

3. Secondary Outcome: Psoriasis Treatment Convenience Scale
Description: Subject assessment of treatment convenience using a Psoriasis Treatment Convenience Scale is defined as a sum of questions 1-5, where each question is scored on a scale from 1-10.
  How easy was the treatment to apply to the skin? "Very difficult" is 1 and "Very easy" is 10 How greasy was the treatment when applying it to the skin? "Very greasy" is 1 and "Not greasy" is 10 How moisturised did your skin feel after applying the treatment? "Not moisturized" is 1 and "Very moisturized" is 10 How greasy did your skin feel after applying the treatment? "Very greasy" is 1 and "Not greasy" is 10 How much did treating your skin disrupt your daily routine? "Very disturbing" is 1 and "Not disturbing" is 10
Time Frame: 8 weeks
Population: The analysis population is defined as those patients from the PP population that have used study medication within 7 days prior to the day of assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Vehicle
Number analyzed (Participants) | 295 | 275 | 87
score on a scale | 41.6 (6.6) | 37.8 (7.6) | 37.2 (7.1)

ADVERSE EVENTS:
Time Frame: AEs were collected/assessed during the screening period (up to 4 weeks) and during the 8 weeks treatment period.
Arm/Group | MC2-01 Cream | CAL/BDP Combination | Vehicle
All-Cause Mortality (participants affected / at risk) | 1/342 | 0/337 | 1/115
Serious Adverse Events (participants affected / at risk) | 9/342 | 11/337 | 5/115
Other Adverse Events (participants affected / at risk) | 0/342 | 0/337 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MC2-01 Cream (N=342) | CAL/BDP Combination (N=337) | Vehicle (N=115)
Abscess (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Angina Pectoris (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Renal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Cervical Vertebral Fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Nosocomial infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Application site cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Diverculitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cervix Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Ischaemic stroke (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Death (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less or equal to 60 days from the time submitted to the sponsor for review. At the end of the Review Period, the sponsor may reasonably require that publication be delayed to permit the filing of patent application. Publication shall not be delayed more than 90 days after receipt of the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/99/NCT03308799/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03308799/SAP_001.pdf